CLINICAL TRIAL: NCT05469919
Title: A Phase 1, Open-label Study to Assess the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of Ceralasertib Administered to Japanese Patients With Advanced Solid Malignancies
Brief Title: An Open-Label Phase 1 Study of Ceralasertib in Japanese Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5330C00014
Record Dates: First submitted 2022-05-18; First posted 2022-07-22 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Malignancies
Keywords: Phase 1; Safety; Tolerability; Pharmacokinetics; Advanced solid malignancies
MeSH Terms: interventions — ceralasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ceralasertib monotherapy (Experimental): This is a sequential group treatment/dose-escalation study with 2 cohorts with no masking.
  Interventions: Drug: Ceralasertib

INTERVENTIONS:
Drug: Ceralasertib — Ceralasertib taken orally

SUMMARY:
This is a Phase 1, open-label study designed to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor activity of ceralasertib in Japanese patients with advanced solid malignancies. Cycle 0 duration is 4 days and each cycle from Cycle 1 has a duration of 28 days.

DETAILED DESCRIPTION:
<Objectives>

Primary Objective:

To investigate the safety and tolerability of ceralasertib in Japanese patients with advanced solid malignancies

Secondary Objective:

To assess the anti-tumor activity and efficacy of ceralasertib. To characterize the first- and multiple-dose pharmacokinetics of ceralasertib.

Exploratory Objective:

To conduct exploratory research into factors that may be predictive of response or may influence the progression of cancer and/or response (efficacy, tolerability, or safety) to ceralasertib.

<Overall design> This is a Phase 1, open-label study designed to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor activity of ceralasertib in Japanese patients with advanced solid malignancies. Cycle 0 duration is 4 days and each cycle from Cycle 1 has a duration of 28 days.

Ceralasertib 240 mg monotherapy in cohort 1 will be orally administered as a single dose at Cycle 0 (Cycle 0 duration is 4 days) Day 1 and twice daily from Day 1 to Day 7 of each 28-day cycle (from Cycle 1). Ceralasertib monotherapy of 160 mg will be orally administered as a single dose at Cycle 0 (Cycle 0 duration is 4 days) Day 1 and twice daily from Day 1 to Day 14 of each 28-day cycle (from Cycle 1), respectively, in cohort 2. Each patient will undergo an DLT evaluation period (Cycle 0 and 1) to have the DLT of ceralasertib determined. Patients will continue with the treatment until disease progression, unacceptable toxicity, or withdrawal from the study.

A minimum of 3 and a maximum of 6 evaluable patients will be enrolled in each cohort ("rolling 6 design"). If no DLT is observed in 3-6 evaluable patients or only 1 DLT is observed in 6 evaluable patients in the current cohort, then transition to the following cohort may occur. If 2 or more patients experience a DLT in each cohort of up to 6 evaluable patients, irrespective of the number of patients enrolled, the dose will be considered not tolerated and recruitment to the current cohort and transition to the following cohort will cease. At the completion of the current cohort, a decision will be made to begin the following cohort based on the SRC review. If no DLT is observed in a 3-6 evaluable patients or only 1 DLT is observed in 6 evaluable patients in a dose setting, the dose is considered tolerated.

Other doses/schedules/combination or cohort expansion may be implemented based on emerging data and the SRC review.

ELIGIBILITY:
Major Inclusion Criteria:

1. Signed written informed consent.
2. At least 18 years of age at the time of signing the ICF.
3. Histological or cytological confirmation of a solid, malignant tumor that is refractory to standard therapies or for which no standard therapies exist.

   Measurable or non-measurable disease according to RECIST version 1.1.
4. Eastern Cooperative Oncology Group/World Health Organization (ECOG/WHO) performance status of 0 to 1 with no deterioration between screening and the first dose of the study treatment, and a minimum life expectancy of 12 weeks
5. Body weight >30 kg and no cancer-associated cachexia (e.g., common terminology criteria for adverse events [CTCAE] Grade 2 or worse weight loss over the past 3 months).

Major Exclusion Criteria:

1. History of another primary malignancy except for:

   * Malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of the study drug and of low potential risk for recurrence
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   * Adequately treated carcinoma in situ without evidence of disease
2. Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting the study treatment, with the exception of alopecia and chemotherapy-related peripheral neuropathy.
3. Presence of life-threatening metastatic visceral disease, as judged by the investigator, uncontrolled central nervous system (CNS) metastatic disease. Patients with spinal cord compression and/or brain metastases may be enrolled if definitively treated (e.g., surgery or radiotherapy) and stable off steroids for at least 4 weeks prior to start of the study treatment.
4. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (known positive hepatitis B virus [HBV], surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies).

   Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if the polymerase chain reaction is negative for HCV RNA.
5. Diagnosis of ataxia telangiectasia.
6. Refractory nausea and vomiting, chronic gastrointestinal diseases, or previous significant stomach/bowel resection, with clinically significant sequelae that would preclude adequate dissolution/absorption of ceralasertib. Partial gastrectomy with preservation of gastric pyloric function and partial resection of the large intestine can be eligible, but inclusion of patients with gastric pylorus resection or patients with duodenum, jejunum or ileum resection requires discussion with the sponsor.
7. Past medical history of interstitial lung disease (ILD) / pneumonitis requiring steroid treatment or any evidence of clinically active ILD / pneumonitis or potential ILD / pneumonitis which is not excluded by the screening test.
8. Treatment with any of the following:

   1. Any investigational medicinal product or other systemic anticancer treatment within 4 weeks prior to the first dose of the study treatment, except for immunotherapy or antibody therapy which has five-fold half-life >4 weeks is within 8 weeks.

      Note: androgen-deprivation therapy is permitted for patients with prostate cancer
   2. The potent inducers or inhibitors of CYP3A within 2 weeks of the first dose of the study treatment; except for St. John's wort, which is 3 weeks.
   3. Prior exposure to an ATR inhibitor.
   4. Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of the study treatment
   5. Radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of the study treatment.
9. Participation in any clinical research study involving treatment with any investigational drug, radiotherapy or surgery, except for the non-treatment phases of these studies, e.g., follow-up phase.
10. History of hypersensitivity to active or inactive excipients of ceralasertib or drugs with a similar chemical structure or class to ceralasertib.
11. Patient has any of the following cardiac criteria:

    1. Mean QT interval corrected by Fridericia's formula (QTcF) for heart rate ≥470 ms calculated from ECGs.
    2. Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG, e.g., complete left bundle branch block, third degree heart block, second degree heart block, first degree heart block.
    3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval.
    4. Patients with uncontrolled hypertension-blood pressure (BP) ≥150/95 mmHg despite medical therapy.
    5. Patients with relative hypotension (BP<100/60 mmHg) or clinically relevant orthostatic hypotension, including a fall in blood pressure of >20 mmHg.
    6. Unstable atrial fibrillation or unstable cardiac arrhythmia with a ventricular rate >100 bpm on an ECG at rest.
    7. Symptomatic heart failure-New York Heart Association Grade II to Grade IV.
    8. Prior or current cardiomyopathy.
    9. Severe valvular heart disease.
    10. Uncontrolled angina (Canadian Cardiovascular Society Grade II to Grade IV despite medical therapy) or acute coronary syndrome within 6 months prior to screening.
    11. Patients at risk of brain perfusion problems, e.g., carotid stenosis. Stroke or transient ischemic attack in the last 6 months prior to screening.
12. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values. Note that growth factor or blood transfusion support to solely meet the criteria is prohibited for 14 days prior to the screening test unless otherwise noted:

    1. Absolute neutrophil count [ANC] <1.5 × 109/L.
    2. Platelet count <100 × 109/L.
    3. Haemoglobin <9 g/dL with no blood transfusions (packed red blood cells) in the past 28 days.
    4. Persisting (>4 weeks) severe pancytopenia due to previous therapy rather than disease (ANC <1.5 × 109/L or platelets <100 × 109/L).
    5. Alanine aminotransferase (ALT) >2.5 × the upper limit of normal (ULN).
    6. Aspartate aminotransferase (AST) >2.5 × ULN.
    7. Total bilirubin (TBL) >1.5 × ULN or >3 × ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia).
    8. Alkaline phosphatase (ALP) >2.5 × ULN (and liver disease unrelated to the tumor).

       Patients with elevated ALP due to tumor related bone metastases or liver metastases will be eligible.
    9. Creatinine clearance <45 mL/min calculated by Cockcroft-Gault equation
    10. Haematuria: +++ on microscopy or dipstick.
    11. INR ≥1.5 or other evidence of impaired hepatic synthesis function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
The number of subjects with dose-limiting toxicity, as defined in the protocol. | From the first dose of study treatment Up to and including the end of cycle 1(each cycle is 28 days).
  Dose-limiting toxicity as described in the protocol that is not related to disease progression, intercurrent illness or concomitant medications and that, despite optional therapeutic intervention, meets protocol-defined criteria.
Safety and tolerability in terms of adverse events | From the first dose of study treatment until 28 days after the last dose.
  Number of subjects with adverse events as a measure of safety and tolerability including changes in vital signs, electrocardiograms (ECGs), safety and laboratory parameters

SECONDARY OUTCOMES:
Overall response rate | At screening and Every 8 weeks ±1 week relative to the start of therapy (Cycle 1 Day 1, each cycle is 28days) until objective disease progression as defined by RECIST version 1.1
  Antitumor activity by evaluation of tumor response assessments using RECIST 1.1
Duration of Response | At screening and Every 8 weeks ±1 week relative to the start of therapy (Cycle 1 Day 1, each cycle is 28 days) until objective disease progression as defined by RECIST version 1.1
  Antitumor activity by evaluation of tumor response assessments using RECIST 1.1
Percentage Change in Tumour Size | At screening and Every 8 weeks ±1 week relative to the start of therapy (Cycle 1 Day 1, each cycle is 28 days) until objective disease progression as defined by RECIST version 1.1
  Antitumor activity by evaluation of tumor response assessments using RECIST 1.1
Progression Free Survival | From start of treatment until the date of objective disease progression or death. (approximately 6 months).
  Antitumor activity by evaluation of tumor response assessments using RECIST 1.1
Plasma ceralasertib concentration(Cmax) | Cycle 0 Day1 to Day4, Cycle1 Day1 and Cycle 1 Day 7 or Day 8. At the end of Cycle1(each cycle is 28 days)
  Observed PK parameters of ceralasertib
Area under the plasma concentration versus time curve(AUC) | Cycle 0 Day1 to Day4, Cycle1 Day1 and Cycle1 Day7 or Day8. At the end of Cycle1(each cycle is 28 days)
  Observed PK parameters of ceralasertib.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Chūōku, Japan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Kuboki Y, Matsubara N, Nakajima H, Fujisawa T, Koyama T, Sato J, Katsuya Y, Kmieciak A, Slade D, Iwata K, Takahashi Y, Nii M, Murayama K, Kawata T, Kawasumi H, Yamamoto N. Ceralasertib, an ATR kinase inhibitor, as monotherapy in Japanese patients with advanced solid malignancies: Results from a phase 1 study. Invest New Drugs. 2025 Dec;43(6):1235-1246. doi: 10.1007/s10637-025-01592-x. Epub 2025 Dec 6. PMID 41351730